CLINICAL TRIAL: NCT00005179
Title: Diet, Exercise and Cardiovascular Health Among Ethnic Children
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1057; R03HL047534 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2000-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

SUMMARY:
To document the patterns of influence or socialization from parents to children in regard to the transmission of cardiovascular disease risk related behaviors such as diet and physical activity.

DETAILED DESCRIPTION:
BACKGROUND:

While much of the research in heart disease prevention has focused on relationships among cardiovascular disease risk factors, cardiovascular disease morbidity and mortality, there is a growing recognition of the importance of various health behaviors, such as what people eat, how much they exercise, if they smoke, their habitual approach to life including Type A behavior. Many of these risk related behaviors are correlated with the various cardiovascular disease risks. This study determined differences in social influence patterns in regard to diet and exercise between obese and non-obese families, and the impact on the obesity, dietary and exercise habits, and risk factors of children beginning at three to four years of age until seven to eight years.

DESIGN NARRATIVE:

This prospective, longitudinal study collected data on the twelve cohorts of families. Blood pressures, resting pulse, height, weight, skinfolds, plasma cholesterol fractions and Type A behavior data were collected on the children at five times over the course of five years. During the four years between each of the clinic measurements, observational data were collected on the diet and exercise habits of the children. At the time of clinic assessment, clinic data were also collected on the parents of the children and self report data on the parents' diet, exercise habits, and other psychosocial variables. Two substudies were also conducted. The first assessed energy expenditure levels of children in the three age groups of 3-4 years, 5-6 years, and 7-8 years and the three body types of lean, average, and obese in 12 different activities. The second substudy assessed the accuracy of mothers' 24-hour recall of the diet and exercise behaviors of their 3-4 year old children as compared to observational data on the same behaviors.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1985-09; Study Completion 1990-06

REFERENCES:
- [Background] Baranowski T, Hooks P, Tsong Y, Cieslik C, Nader PR. Aerobic physical activity among third- to sixth-grade children. J Dev Behav Pediatr. 1987 Aug;8(4):203-6. PMID 3611360
- [Background] Eck LH, Klesges RC, Hanson CL, Baranowski T, Henske J. A comparison of four commonly used nutrient database programs. J Am Diet Assoc. 1988 May;88(5):602-4. PMID 3367021
- [Background] Hooks PC, Tsong Y, Baranowski T, Henske JC, Nader PR, Levin JS. Recruitment strategies for multiethnic family and community health research. Fam Community Health. 1988 May;11(1):48-59. doi: 10.1097/00003727-198805000-00009. No abstract available. PMID 10286764
- [Background] Baranowski T, Tsong Y, Henske J, Dunn JK, Hooks P. Ethnic variation in blood pressure among preadolescent children. Pediatr Res. 1988 Mar;23(3):270-4. doi: 10.1203/00006450-198803000-00008. PMID 3353173
- [Background] Brodwick M, Baranowski T, Rassin DK. Patterns of infant feeding in a tri-ethnic population. J Am Diet Assoc. 1989 Aug;89(8):1129-32. No abstract available. PMID 2760374
- [Background] Baranowski T, Bryan GT, Rassin DK, Harrison JA, Henske JC. Ethnicity, infant-feeding practices, and childhood adiposity. J Dev Behav Pediatr. 1990 Oct;11(5):234-9. PMID 2258441
- [Background] Baranowski T, Tsong Y, Brodwick M. Scaling of response scale adverbs among black-American adults. Percept Mot Skills. 1990 Oct;71(2):547-59. doi: 10.2466/pms.1990.71.2.547. PMID 2251088
- [Background] Baranowski T: Validity of Self Report of Physical Activity: An Information Processing Approach. Research Quarterly for Exercise and Sport, (in press), 0000
- [Background] Perry C, Baranowski T, Parcel G: Social and Environmental Triggers and Reinforcements for Health Behavior: Social Learning Theory. In: Glanz K, Lewis FM, Rimer B, (Eds) Health Behaviors and Health Education Theory, Research and Practice. San Francisco: Jossey-Bass, (in press), 0000
- [Background] Baranowski T, Bryan GT, Harrison JA, Rassin DK, Greaves KA, Baranowski JH. Height, infant-feeding practices and cardiovascular functioning among 3 or 4 year old children in three ethnic groups. J Clin Epidemiol. 1992 May;45(5):513-8. doi: 10.1016/0895-4356(92)90100-2. PMID 1588357
- [Background] Higginbotham JC, Baranowski T, Puhl J, Greaves KA. Ethnicity, gender, and Type A differences in resting heart rate and blood pressure among young children. Ethn Dis. 1991 Spring;1(2):123-34. PMID 1842529
- [Background] Treiber FA, Baranowski T, Braden DS, Strong WB, Levy M, Knox W. Social support for exercise: relationship to physical activity in young adults. Prev Med. 1991 Nov;20(6):737-50. doi: 10.1016/0091-7435(91)90068-f. PMID 1766945
- [Background] Baranowski T, Sprague D, Baranowski JH, Harrison JA. Accuracy of maternal dietary recall for preschool children. J Am Diet Assoc. 1991 Jun;91(6):669-74. PMID 2040780
- [Background] Durant RH, Baranowski T, Davis H, Thompson WO, Puhl J, Greaves KA, Rhodes T. Reliability and variability of heart rate monitoring in 3-, 4-, or 5-yr-old children. Med Sci Sports Exerc. 1992 Feb;24(2):265-71. PMID 1549018
- [Background] Puhl J, Greaves K, Hoyt M, Baranowski T. Children's Activity Rating Scale (CARS): description and calibration. Res Q Exerc Sport. 1990 Mar;61(1):26-36. doi: 10.1080/02701367.1990.10607475. PMID 2091164
- [Background] DuRant RH, Baranowski T, Puhl J, Rhodes T, Davis H, Greaves KA, Thompson WO. Evaluation of the Children's Activity Rating Scale (CARS) in young children. Med Sci Sports Exerc. 1993 Dec;25(12):1415-21. PMID 8107551
- [Background] Baranowski T, Domel SB. A cognitive model of children's reporting of food intake. Am J Clin Nutr. 1994 Jan;59(1 Suppl):212S-217S. doi: 10.1093/ajcn/59.1.212S. PMID 8279427
- [Background] Baranowski T, Thompson WO, DuRant RH, Baranowski J, Puhl J. Observations on physical activity in physical locations: age, gender, ethnicity, and month effects. Res Q Exerc Sport. 1993 Jun;64(2):127-33. doi: 10.1080/02701367.1993.10608789. PMID 8341835